CLINICAL TRIAL: NCT06285227
Title: A Randomized, Open/Double-blind, Placebo-controlled Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of CM313 in Healthy Subjects With Single Subcutaneous Injection/Intravenous Infusion
Brief Title: Study of CM313 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM313-100001
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): CM313, subcutaneous injection, once
  Interventions: Biological: CM313 injection
- Group 2 (Experimental): CM313, subcutaneous injection, once
  Interventions: Biological: CM313 injection
- Group 3 (Experimental): CM313, subcutaneous injection, once
  Interventions: Biological: CM313 injection
- Group 4 (Experimental): CM313, infusion, once
  Interventions: Biological: CM313 injection

INTERVENTIONS:
Biological: CM313 injection — CM313

SUMMARY:
This study is a single center, randomized, open/double-blind, placebo-controlled, single dose, dose escalation Phase I clinical study aimed at evaluating the safety, tolerability, pharmacokinetics, pharmacokinetic characteristics, and immunogenicity of CM313 administered subcutaneously or intravenously at different doses in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age ≥ 18 years & ≤50 years.
* Subjects voluntarily signed the Informed Consent Form and were able to comply with the provisions of this protocol.

Exclusion Criteria:

* With history of malignant tumors;
* Plan to undergo major surgery during the research period
* Known to be allergic to monoclonal antibody drugs or other related drugs, food, or CM313 excipients;
* With any voluntary blood donation or any other form of blood loss exceeding 400 mL;
* The average daily smoking volume within the first three months of screening is greater than 5 cigarettes;
* Positive results in baseline alcohol breath test or urine drug abuse screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event | Up to week 12
  Incidence, severity, and outcome of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhang, Principal Investigator — Huashan Hospital; Yu Xue, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, China

REFERENCES:
- [Derived] Yu S, Wu J, Zhao J, He J, Yan H, Zhang X, Yang Y, Song H, Hou Q, Guo B, Qiu Y, Chen B, Xue Y, Zhang J. Pharmacokinetics, Pharmacodynamics, and Immunogenicity of CM313 in Healthy Participants: An Open-Label/Double-Blind, Randomized, Placebo-Controlled Phase 1 Trial. Clin Transl Sci. 2025 Sep;18(9):e70334. doi: 10.1111/cts.70334. PMID 40965985